CLINICAL TRIAL: NCT00344448
Title: A Randomized, Placebo Controlled, Proof of Concept, Study of Raptiva, a Humanized Anti-CD-11a Monoclonal Antibody, in Patients With Sjogren's Syndrome
Brief Title: Pilot Study of Raptiva to Treat Sjogren's Syndrome
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Increased risk of PML associated with raptiva in other studies
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Principal Investigator, Gabor Illei, M.D., Head of Sjogren's Syndrome Clinic, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 060181; 06-D-0181 (Other: The National Institutes of Health)
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Results first posted 2015-12-21 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Sjogren's Syndrome
Keywords: Adhesion Molecule; Interventional Study; Immunomodulation; Autoimmunity; Sjogren Syndrome; SS
MeSH Terms: conditions — Sjogren's Syndrome; Autoimmune Diseases | interventions — efalizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Raptiva (Experimental): At the beginning of the first (week 1) and second (week 13) phases, all patients will receive reduced dose of the study medication determined at 0.7 mg/kg/week. During all the subsequent administrations, all patients will receive full dose of the study medication determined at 1 mg/kg/week.
  Interventions: Drug: Raptiva
- placebo (Placebo Comparator): Weekly subcutaneous injection of a placebo (formulated to match the commercial vial of Raptiva in appearance and content except for the active ingredient) for the first 12 weeks of the study.
  Interventions: Drug: Raptiva

INTERVENTIONS:
Drug: Raptiva — During the first phase of the study, subjects are randomized in a double blind fashion to receive weekly subcutaneous injections of efalizumab (Raptiva) or placebo (weeks 0-12). The second 12 weeks long phase is open label with all subjects receiving weekly subcutaneous injections of efalizumab.
  Other Names: efalizumab; anti-CD11a monoclonal antibody

SUMMARY:
This study will examine the effect of the drug Raptiva (efalizumab) in patients with Sjögren's syndrome (SS), an autoimmune disease affecting the glands producing saliva & tears. The cause of SS is not known, but inflammation plays an important role. Raptiva is approved by the Food and Drug Administration to treat psoriasis, an inflammatory skin disease. Patients 18 years of age & older with SS may be eligible for this study. Candidates are screened with a history & physical examination, chest x-ray, and oral & eye examinations.

Participants are randomly assigned to receive either Raptiva or placebo (an inactive substance that looks like Raptiva) for the first 3 months of the study. For the next 3 months, all participants receive Raptiva. Both Raptiva & placebo are injected under the skin once a week. Evaluation during treatment & for 2 months after treatment as follows:

Full comprehensive evaluations (beginning of the study, at weeks 13 & 25 and 2 months after treatment ends):

* Physical examination & blood draw.
* Saliva collection done in two ways: 1) suctions cups connected to collection tubes are placed over the salivary gland ducts in the mouth and under the tongue; and 2) a sour-tasting liquid is applied to the top & sides of the tongue at 30-second intervals to stimulate saliva production.
* Eye exam for tear gland function.
* Questionnaires about mouth & eye dryness, energy level and overall well-being.
* Lip biopsy (screening & week 13 visits only). A few minor salivary glands are removed for examination under a microscope. The lower lip is numbed, a small cut is made on the inside of the lip, and several glands are removed. The cut is closed with a few stitches that are removed after 5 to 7 days.
* Magnetic resonance imaging of the parotid glands (salivary glands near the ear) at weeks 1, 13 and 25. The patient lies on a stretcher that is moved into the scanner (a metal cylinder containing a strong magnetic field). The head is held in place during the scan. The study lasts about 90 minutes.
* Short evaluations at weeks 3, 5, 9, 15, 17, 21 and 1 month after treatment ends.
* Medical history & physical examination, blood draw, evaluation for changes in symptoms and side effects, review of current medications at weeks 3, 9, 15 and 21.
* Laboratory tests, evaluation for changes in symptoms and side effects, review of current medications, saliva collection without the sour liquid and short evaluation of tear production at weeks 5 and 17.
* Blood tests at week 29

DETAILED DESCRIPTION:
The LFA-1/ICAM-1 interaction is important in migration of lymphocytes to inflammatory sites, T-lymphocyte activation, antigen presentation, and maintaining the integrity of the immunologic synapse. In both murine and human Sjogren's Syndrome, increased expression of LFA-1 was found on activated lymphocytes, and increased expression of ICAM-1 was present on the activated endothelial cells in the diseased salivary and lacrimal glands. In animal models, blockade of the LFA-1/ICAM-1 interaction resulted in reduction of glandular inflammation.

Raptiva (efalizumab) is a recombinant humanized monoclonal antibody that binds to human CD11a, the alpha-subunit of Leukocyte Function Antigen-1 (LFA-1) and inhibits the LFA-1/ICAM-1 interaction. Raptiva is an FDA-approved medication for treatment of mild-to-moderate psoriasis.

In this pilot, proof of concept, randomized, double-blind, placebo-controlled study, up to 25 patients with Sjogren's syndrome may be enrolled. In the first, double-blind phase of the study, patients will be randomized and treated with weekly subcutaneous (SC) injections of either Raptiva (1mg/kg) or placebo for 12 weeks. In the second open label phase, all patients will be treated with weekly SC injections of Raptiva (1mg/kg) for another 12 weeks and then followed for an additional 8 weeks. Safety will be evaluated using standard clinical and laboratory parameters. To assess the potential effect of Raptiva on Sjogren's syndrome, minor salivary gland biopsy, oral and ocular evaluations, and measurements of surrogate markers of inflammation will be compared between the Raptiva and placebo treated groups before and after the treatment. Patients who either do not tolerate the drug or have worsening in their disease activity will be withdrawn from the protocol.

If Raptiva is well tolerated in this study and the treatment is associated with improvement in clinical parameters of Sjogren's Syndrome, further large studies of efficacy are planned.

ELIGIBILITY:
* INCLUSION CRITERIA:

Up to 25 patients may be enrolled in this study to obtain at least 20 patients to complete the study and to allow for an estimated up to 20% early attrition rate. Eligible patients will have primary SS diagnosed according to the American-European Consensus Group Sjogren's Syndrome Classification Criteria. Subjects will be chosen based on their potential capacity to reverse the inflammatory process and at least partially recover the exocrine function in the salivary and lacrimal glands, as indicated in the inclusion criteria by requiring a minimal level of salivary flow as a marker of functional gland tissue. Pre-screening, which would include ophthalmologic evaluation, standard laboratory tests, and minor salivary gland biopsy, will be performed under the natural history protocol, and eligible patients will be offered to sign the informed consent for this protocol.

Age at entry at least 18 years

Must give written informed consent prior to entry in the protocol.

Must fulfill at least 4 of the 6 following criteria for Primary SS as defined by the American-European Consensus Group Sjogren's Syndrome Classification Criteria, including either item IV or VI, or fulfill 3 of the 4 objective criteria (III, IV, V, VI) [53] :

Ocular symptoms (at least one):

Dry eyes greater than 3 months

Foreign body sensation in the eyes

Use of artificial tears greater than 3x/day

Oral symptoms (at least one):

Dry mouth greater than 3 months

Swollen salivary glands

Need liquids to swallow dry foods

Ocular signs (at least one):

Schirmer test (without anesthesia) less than or equal to 5 mm/5 min

Positive vital dye staining (van Bijsterveld greater than or equal to 4)

Histopathology: Minor salivary gland biopsy showing focal lymphocyte sialoadenitis (focus score greater than or equal to 1 per 4 mm(2))

Oral signs (at least one):

Unstimulated whole salivary flow (less than or equal to 1.5 ml in 15 min)

Abnormal parotid sialography

Abnormal salivary scintigraphy

Autoantibodies (at least one):

Anti-SSA or Anti-SSB

One or more of the following:

Serum ANA level greater than or equal to 1EU

Serum Anti-SSA level greater than or equal to 20EU

Serum Anti-SSB level greater than or equal to 20EU

Serum RF level greater than or equal to 20 IU/ml

One or more of the following:

ESR greater than 25 mm/hr for men; ESR greater than 42 mm/hr for women

Serum IgG level greater than or equal to 1750 mg/dl

Serum CRP level greater than or equal to 0.8 mg/dl

Stimulated salivary flow of at least 0.1 ml/min.

Minor salivary gland biopsy with a focus score of greater than or equal to 4 within at most 12 months prior to the study enrollment.

Score of 3 or more on Oxford scale in at least one eye at the study entry.

Negative age- and gender- appropriate malignancy screening for breast, cervical, colorectal cancer for women; and prostate and colorectal cancer for men. Specifically:

* All women: pelvic exam with Papanicolaou smear within one year of study entry.
* Women age 40 and older: mammogram within 1 year of study entry,
* Both genders age 50 and older; stool screening for occult blood within one year, or flexible sigmoidoscopy or colonoscopy within five years
* Men age 50 and older: rectal examination or prostate specific antigen testing

EXCLUSION CRITERIA:

Past head and neck irradiation.

Hepatitis B, C, HIV, or HTLV infection.

History of lymphoma or monoclonal gammopathy of unknown significance (MGUS).

Sarcoidosis.

Graft-versus-host disease.

Women of childbearing potential are required to have a negative pregnancy test at screening.

Women of childbearing potential and fertile men who are not practicing or who are unwilling to practice birth control during and for a period of three months after the completion of the study.

Any therapy with human or murine antibodies or any experimental therapy within 3 months.

Therapy with cyclophosphamide, pulse methylprednisolone or IVIg, azathioprine, mycophenolate mofetil, oral cyclosporine or methotrexate within 4 weeks of first study treatment.

History of rituximab therapy.

Prednisone dose greater than or equal to 10 mg/day.

Allergy to murine or human antibodies.

History of anaphylaxis.

Serum creatinine greater than 2.0 mg/dl.

History of any malignancy.

Active infection that requires the use of intravenous antibiotics and does not resolve within 1 week of Day 1.

Any active viral infection that does not resolve within 10 days prior to Day 1.

WBC less than 2000/microL or ANC less than 1500/microL or Hgb less than 9.0 g/dL or platelets less than 150,000/microL or absolute lymphocyte count less than or equal to 500/microL.

ALT and/or AST greater than 1.5x upper limit of normal (ULN) or alkaline phosphatase greater than 1.5x ULN.

Significant concurrent medical condition that, in the opinion of the Principal Investigator, could affect the patient's ability to tolerate or complete the study.

Live vaccines within 12 weeks of first treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-06; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gabor G Illei, MD, PhD, MHS, Principal Investigator — National Institute of Dental and Craniofacial Research (NIDCR)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Skopouli FN, Moutsopoulos HM. Autoimmune epitheliitis: Sjogren's syndrome. Clin Exp Rheumatol. 1994 Nov-Dec;12 Suppl 11:S9-11. PMID 7768059
- [Background] Atkinson JC, Fox PC. Sjogren's syndrome: oral and dental considerations. J Am Dent Assoc. 1993 Mar;124(3):74-6, 78-82, 84-6. doi: 10.14219/jada.archive.1993.0064. PMID 8335784
- [Background] Garcia-Carrasco M, Ramos-Casals M, Rosas J, Pallares L, Calvo-Alen J, Cervera R, Font J, Ingelmo M. Primary Sjogren syndrome: clinical and immunologic disease patterns in a cohort of 400 patients. Medicine (Baltimore). 2002 Jul;81(4):270-80. doi: 10.1097/00005792-200207000-00003. No abstract available. PMID 12169882
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/detail/B_2006-D-0181.html

RESULTS

PARTICIPANT FLOW:
Period: Screening
Arm/Group | Raptiva | Placebo
Started | 6 (No randomization during the screening phase) | 4
Completed | 6 | 3
Not Completed | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Double Blind, Placebo Controlled
Arm/Group | Raptiva | Placebo
Started | 6 | 3
Completed | 4 | 3
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Study terminated | 1 | 0
Period: Open Label
Arm/Group | Raptiva | Placebo
Started | 4 | 3
Completed | 2 | 2
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Study terminated | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Raptiva | Placebo | Total
Number analyzed (Participants) | 6 | 3 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 3 | 9
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 51 (13.3) | 53 (4.16) | 53 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 | 8
  Male | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 6 | 3 | 9

OUTCOME MEASURES:

1. Primary Outcome: Response Rate at the End of the First (Blinded, Placebo Controlled) Phase at 12 Weeks
Description: Patient will be considered a responder if (s)he demonstrates improvement in 2 / 3 disease activity measures without worsening of the third one.
  1. Salivary flow: 0.45 ml / 15 min improvement in unstimulated whole salivary flow from baseline value obtained at the study entry.
  2. Salivary gland biopsy:
     at least 2 points improvement in the focus score on MSG biopsy
  3. Tear flow:
  at least 30% improvement in ophthalmic Oxford grading scheme or normalization of the scale as defined by score of 0 or 2mm improvement in Schirmer test as compared with the baseline in either eye.
Time Frame: 3 months
Measure: Number; unit: participant
Arm/Group | Raptiva | Placebo
Number analyzed (Participants) | 6 | 3
participant | 0 | 1

ADVERSE EVENTS:
Time Frame: 2 years and 5 month
Description: Raptiva: AEs occuring in 6 patients receiving Raptiva durig the blinded phase plus the 2 patients who received placebo during the blinded phase but received Raptiva during the open lable phase.
  Placebo AEs occuring in the placebo group (n=3) during the blinded phase. One patient withdrew after completing the placebo phase.
Arm/Group | Raptiva | Placebo
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 8/8 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Raptiva (N=8) | Placebo (N=3)
Angular cheilitis (Infections and infestations) | 0 (0) | 1 (1)
Corneal scratches (Eye disorders) | 2 (2) | 1 (1) — Traumatic
Diarrhea (Gastrointestinal disorders) | 1 (1) | 2 (5)
Dysuria (Renal and urinary disorders) | 2 (2) | 0 (0)
Flulikr symptoms (General disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Increase in autoantibody titers (Immune system disorders) | 2 (2) | 1 (1)
Increased sweating (General disorders) | 1 (1) | 0 (0)
Infectious parotitis (Infections and infestations) | 1 (1) | 0 (0)
Keratoconjunctivitis (Eye disorders) | 2 (2) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Monoclonal gammopathy (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — M-spike on immunefixation electrophoresis
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oral ulcers (Infections and infestations) | 6 (7) | 1 (1)
Pleuritic chest pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Sinusitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Tooth abscess (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 1 (1)
Vaginal dryness (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Vaginal yeast infection (Infections and infestations) | 1 (1) | 1 (1)
right upper quadrant pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0)
Oligoclonal gammopathy (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
oral candidiasis (Infections and infestations) | 2 (2) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Parotid pain (General disorders) | 1 (1) | 0 (0) — on citric acid stimulation
Parotitis (Metabolism and nutrition disorders) | 3 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination due to serious adverse event described in psoriasis which led to the withdrawal of the drug from market.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes